CLINICAL TRIAL: NCT04456985
Title: Effect of Preoperative Intervention With Folic Acid and Vitamin B12 on Postoperative Neurobehavioral Changes in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Zhang Lei, Deputy Chief Physician and Associate Researcher, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SH9H-2020-T57-2
Record Dates: First submitted 2020-06-14; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Folic Acid; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Before the operation, the patient took 20ml of brown sugar aqueous solution containing folic acid and VitB12 for 3 days (folic acid concentration is 0.4mg / d for 2 year old children + 1.2μg / d of VitB12, dissolved in 20ml brown sugar water once a day). Postoperatively, PAED scores were performed at the time of awakening, extubation and every 10min within 30min after extubation. 10 points is defined as delirium during the recovery period). Long-term neurobehavioral changes were evaluated using the Gesell scale, followed up every six months until the age of three
  Interventions: Dietary Supplement: Folic acid and vitamin B12
- Placebo group (Placebo Comparator): The patients in the placebo group took 20 ml of brown sugar aqueous solution with the same concentration as the intervention group 3 days before the operation. Postoperatively, PAED scores were performed at the time of recovery, extubation, and every 10 minutes within 30 minutes after extubation. The PAED scores of all children were measured by the same person. (The total score is 0-20, and the score ≥10 is defined as delirium during the recovery period). Long-term neurobehavioral changes were evaluated using the Gesell scale, followed up every six months until the age of three
  Interventions: Dietary Supplement: brown sugar aqueous

INTERVENTIONS:
Dietary Supplement: Folic acid and vitamin B12 — Take folic acid and VitB12 for 3 consecutive days before surgery
  Arms: Intervention group
Dietary Supplement: brown sugar aqueous — take 20 ml of brown sugar aqueous solution with the same concentration as the intervention group 3 days before the operation
  Arms: Placebo group

SUMMARY:
Comparison of preoperative folic acid and VitB12 intervention on postoperative delirium and long-term neurobehavioral changes in children under general anesthesia

DETAILED DESCRIPTION:
Folic acid, as a one-carbon unit transferase coenzyme, participates in the synthesis of purine and thymine, and is an important element of the nervous system. Vitamin B12 participates in methyl conversion and folate metabolism in the body, promoting the conversion of 5-methyltetrahydrofolate to tetrahydrofolate. It has been reported that the lack of serum folic acid and B12 is associated with an increased risk of cognitive impairment. The explanation mechanism of the relationship between folic acid deficiency and cognitive dysfunction may be that folic acid deficiency leads to impaired central nervous system methylation, resulting in insufficient methyl synthesis of myelin sheaths, neurotransmitters, membrane phospholipids and deoxyribonucleic acid. Our previous studies showed that preoperative folic acid supplementation can alleviate myelin damage and cognitive impairment in young rats caused by sevoflurane anesthesia. Therefore, this study further explored the preoperative folic acid and coenzyme B12 supplementation for children's delirium and long-term neurobehavioral changes after general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. ASA grade is Ⅰ ~ Ⅱ;
2. Children aged 6 months to 2 years old;
3. It is planned to undergo head, neck and maxillofacial surgery under general anesthesia with anesthesia for less than 6 hours

Exclusion Criteria:

1. Children with a history of respiratory tract infection within 1 week;
2. Children with congenital malformations such as congenital heart disease;
3. Children with central nervous system diseases or mental disorders or mental disorders;
4. Children with long-term use of sedative or analgesic drugs;
5. Children with severe liver and kidney dysfunction;
6. Received folic acid and VitB12 supplement treatment or taken related derivatives;
7. Have taken drugs that affect absorption within the past month, such as sulfonamides, aspirin, etc .;
8. Those who have participated in other relevant clinical research in the past 3 months;
9. Children with stunting

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
PAED scale | 10 minutes after surgery
  Observe whether the index will cause delirium during the recovery period.The evaluation range of the PAED scale is 0-20 points, If the score exceeds 10 points, Then it is considered delirium.
Gesell scale | 2 day after surgery
  Through the gesell scale, 5 tests are carried out on children: gross motor ability, fine movement, physical ability, verbal ability, and human ability.The evaluation range of the Gesell scale is 0-100 points. If the score is higher, it means good. If the score is low, it means that the result is not good. If the result is not good, it may be caused by anesthesia, so we conducted this evaluation.

SECONDARY OUTCOMES:
Heart Rate | During the induction period of anesthesia, intubation, and the operation period；immediately after entering the resuscitation room (T1), 5 minutes before extubation (T2), immediately after extubation (T3), and 2 minutes after extubation (T4);
  Observe heart rate through a monitor
Mean Blood Pressure | During the induction period of anesthesia, intubation, and the operation period；immediately after entering the resuscitation room (T1), 5 minutes before extubation (T2), immediately after extubation (T3), and 2 minutes after extubation (T4);
  Observe and calculated mean blood pressure through a monitor
Extubation time | immediately after surgery
  Extubation time
Ramsay sedation score | 10 minutes after extubation
  Ramsay sedation score after recovery, extubation and every 10min within 30min after extubation，Ramsay sedation score is 1-6 points. If the score is 2-4 points，That result is satisfactory, 5-6 points are excessive sedation.
Postoperative pain CHEOPs scores | 20 minutes after extubation
  The postoperative pain CHEOPs scores were taken at the time of extubation and every 10 minutes within 30 minutes after extubation (the total score was less than 6 points, there was no pain, and ≥10 points for corresponding analgesia treatment).
  The total score is 46 points, if the total score is less than 6 points, it is judged as no pain
Narcotic drugs | During the surgery
  The use of narcotic drugs (eg pentazocine, propofol)
Other adverse events during the recovery period | Immediately after the surgery
  Other adverse events during the recovery period (eg nausea and vomiting, bronchospasm, respiratory depression, etc.)
recovery time | immediately after recovery
  recovery time

CONTACTS AND LOCATIONS:
Overall Officials: hong jiang, Doctor, Study Director — Director of Anesthesiology
Locations (1):
- China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT04456985/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT04456985/ICF_001.pdf